CLINICAL TRIAL: NCT04545346
Title: The Potential of a Low Glutamate Diet in Refractory Pediatric Epilepsy Patients
Brief Title: The Potential of a Low Glutamate Diet as a Treatment for Pediatric Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Kathleen Holton, Associate Professor, American University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB- 2019- 240
Record Dates: First submitted 2020-08-26; First posted 2020-09-11 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Epilepsy in Children; Epilepsy in Youth; Randomized Controlled Trial; Refractory Epilepsy; Diet Intervention
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-listed control (No Intervention): Participants continue care as usual. All all medications must be kept constant during the study period, unless medically necessary.
- Low Glutamate diet (Experimental): Participants are put on the low glutamate diet for one month. The low glutamate diet reduces the consumption of free glutamate, while optimizing dietary micronutrient and antioxidant intake.
  Interventions: Other: Low Glutamate diet

INTERVENTIONS:
Other: Low Glutamate diet — Participants will be given extensive online dietary training and assigned to follow the low glutamate diet for one month. The low glutamate diet reduces the consumption of free glutamate, while optimizing dietary micronutrient and antioxidant intake.
  Arms: Low Glutamate diet

SUMMARY:
The study is investigating if following the low glutamate diet for 1 month, as compared to care as usual, can improve seizure frequency, severity, and duration; cognitive functioning; and/or quality of life in children with epilepsy.

DETAILED DESCRIPTION:
Epilepsy is estimated to effect 470,000 children within the U.S. About a third of epilepsy patients are refractory. For these patients, dietary therapy is an alternative option. However, current dietary therapies present issues with compliance, palatability, adverse events, and providing necessary nutrients for brain growth and development during childhood. A dietary option that can improve tolerability, increase compliance, and reduce or eliminate adverse effects, while also optimizing nutrient intake, is critical for the advancement of dietary therapy options in epilepsy.

Glutamate is found in the diet as a flavor enhancer; and is also an important neurotransmitter in the body which mediates seizure activity. Dietary sources of free glutamate are common and include numerous food additives (including many hidden sources) and some items which naturally contain higher amounts of glutamate. The low glutamate diet reduces the consumption of free glutamate, while optimizing dietary micronutrient and antioxidant intake, which can protect against the negative effects caused by high glutamate concentrations in the brain. Additionally, the low glutamate diet is balanced, nutritious and palatable, with no side effects.

The study is investigating if following the low glutamate diet for 1 month can improve seizure frequency, severity, and duration; cognitive functioning; and/or quality of life, in children with epilepsy. Participation in the study will be done virtually and over a 2- or 3- month study period, depending on group randomization. All participants will have the opportunity to undergo dietary training and follow the diet.

ELIGIBILITY:
Inclusion Criteria:

* 4 or more seizures per month
* Willing to keep all medications constant during the study.
* All medications have remained constant for 30 days prior to study enrollment
* Any previously attempted dietary therapies stopped before study enrollment

Exclusion Criteria:

* Known or suspected inborn errors of metabolism
* Non-English speaking households

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Change in seizure frequency | At 1 month post treatment
  All families will keep a seizure diary recording the number of daily seizures. This will be used to accurately determine these variables for the last week, which will be recorded on seizure assessment forms.
Change in seizure severity | At 1 month post treatment
  . During the last week of each study period, families will be asked to complete a seizure assessment form. This will include a subjective rating scale for seizure severity with a minimum score of 0 (not severe) and a maximum score of 10 (very severe).
Change in seizure duration | At 1 month post treatment
  All families will keep a seizure diary recording the duration of seizures. This will be used to accurately determine these variables for the last week, which will be recorded on seizure assessment forms.

SECONDARY OUTCOMES:
The effect of a 1-month low-glutamate diet on quality of life in children with epilepsy. | At 1 month post treatment
  Parents will be asked to complete the Quality of Life in Childhood Epilepsy Questionnaire (QOLCE-55). This 55-question quality of life questionnaire has been validated for children ages 4 and older and is used to assess the participant's cognitive, emotional, social, and physical functioning.
The effect of a 1-month low-glutamate diet on cognitive functioning in children with epilepsy. | At 1 month post treatment
  Cognitive function will be assessed via CNSVS, a computerized neurocognitive testing software.
Examine change in resting state brain waves after 1-month on the low glutamate diet | At 1 month post treatment
  Electroencephalography (EEG) will be offered to all participants. Four minutes of eyes-closed and eyes-open resting state EEG data will be recorded at the end of the baseline, wait-listed control, and active intervention periods in a sound-attenuated, air-conditioned room. Participants will sit in a comfortable chair in front of a computer monitor. For eyes-closed recordings, participants will be instructed to sit as still as possible, while staying relaxed but awake. For eyes-open recordings, participants will be instructed to sit as still as possible and to focus on a fixation point on the screen while keeping blinking to a minimum, if possible. Participants will be monitored to make sure they are complying with condition instructions. Mean power (total power of frequency band/width of frequency band) and relative power (absolute power of frequency band/total power or percent) will be calculated for delta, theta, alpha, beta, gamma, high gamma, and total power.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Holton, MPH, PhD, Principal Investigator — American University
Locations (1):
- American University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarlo GL, Kao A, Holton KF. Investigation of the low glutamate diet as an adjunct treatment for pediatric epilepsy: A pilot randomized controlled trial. Seizure. 2023 Mar;106:138-147. doi: 10.1016/j.seizure.2023.02.013. Epub 2023 Feb 20. PMID 36867910